CLINICAL TRIAL: NCT04593186
Title: Trans-oral Magnifying Endoscopy With Narrow Band Imaging for Screening of Nasopharyngeal Carcinoma
Brief Title: Magnifying NBI for Occult NPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Associate consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CRE-2020.426
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma, Narrow band Imaging, Magnifying endoscopy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Narrow Band Imaging

STUDY DESIGN:
Intervention Model Description: Trans-oral magnifying endoscopy with Narrow Band Imaging assessment of nasopharynx
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans-oral magnifying endoscopy with NBI (Experimental): Transoral magnifying endoscopy with High Definition Upper Endoscope with Narrow Band Imaging enhancement (Olympus GIF-H290Z)
  Interventions: Procedure: Trans-oral magnifying endoscopy with NBI

INTERVENTIONS:
Procedure: Trans-oral magnifying endoscopy with NBI — Endoscopic procedures would be performed by endoscopists with expertise on performing magnifying NBI endoscopy. Topical local anaesthetic will be applied to the oropharynx and nasopharynx. In addition, intravenous sedation by use of Midazolam and Fentanyl would be given. Endoscopes with magnification and NBI function would be used (GF-H290Z, Olympus Medical Corporations, Tokyo, Japan). A soft black hood would be attached to the tip of the endoscope for better focal length adjustment.
  Upon insertion through a mouthpiece, the scope will then be retroflexed into the nasopharynx and the lateral walls into the Fossa of Rosenmuller and the posterior nasopharyngeal wall will be systematically examined with white light and NBI. Target suspicious areas would be examined by use of magnification with the power up to 80X. Biopsy would be taken if suspicious lesion is identified during the procedure.

SUMMARY:
Diagnosis of nasopharyngeal carcinoma (NPC) is currently made by trans-nasal endoscopy and biopsy. The small caliber endoscope provides only a limited view of the nasopharynx and may not be able to provide a thorough assessment of the nasopharynx. The investigators have developed a novel endoscopic approach to access the nasopharynx by using a trans-oral high definition endoscope with magnification and image enhancement function. In this cohort study, we aim to investigate the efficacy of diagnosing NPC by applying the novel technique in a high risk patient group with elevated plasma EBV DNA but with negative screening with conventional trans-nasal endoscopy.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in our region and is the 9th most common cancer in Hong Kong. Traditionally diagnosis has been through a nasoendoscopic examination of the nasopharynx with white light followed by a biopsy of suspicious lesions for a confirmatory diagnosis. However, given the geometry of the anatomy of the nasopharynx, with its inherent crevices and varying amounts of lymphoid tissues, lesions are not always easily identified leading to potential missed lesions. The non-specific aspect of white light also leads to excessive biopsies that are not without risk and of some discomfort to patients. Recent advances in liquid biopsies have also allowed for the detection of earlier and smaller lesions that are not always easily identified on nasoendoscopy but rather are seen on Magnetic Resonance Imaging (MRI).

An alternative imaging technique is the use of Narrow Band Imaging (NBI) to view the vasculature of the mucosa to identify suspicious lesions for pre-malignancy and malignancy that has been popularized in the gastrointestinal tract. In NPC, NBI with the flexible nasoendoscopes has been used in the diagnosis of NPC with varying success. Researchers at Chinese University of Hong Kong has found that in NPC NBI has limitations arising from a lack of consensus on vascular findings on NBI that constitute malignancy, lack of magnification and long focal length of current nasoendoscopes1. Flexible endoscopy using conventional esophago-gastroscopy endoscope (OGD) with NBI and magnification power up to 80x overcome the limitations of current nasoendoscopes. The passage of the endoscope through the mouth and retroflexion at oropharynx could visualize the nasopharynx clearly and detailed assessment is feasible.

Here in this study the investigators will seek to use a trans-oral magnifying endoscopy with NBI and retroflexion into the nasopharynx to view the nasopharynx to evaluate the feasibility in the diagnosis of occult nasopharyngeal carcinoma.

The aim of this study is to investigate the clinical usefulness of trans-oral magnifying endoscopy with NBI as a screening tool for patients at increased risk of nasopharyngeal carcinoma (NPC).

The investigators hypothesize that with the use of magnifying NBI trans-oral endoscopy, the nasopharynx could improve the diagnostic yield of NPC in high risk patients with negative test on conventional investigations. As a result, such endoscopic screening tool could be used routinely to identify early NPC in patients deemed at risk.

Study Design

This study is a prospective single arm study designed to evaluate the diagnostic yield of trans-oral magnifying NBI endoscopic assessment of nasopharynx in patients who are deemed elevated risk of NPC but with negative traditional endoscopic and radiological screening.

In a previous study conducted by the Department of Chemical Pathology and Otorhinolaryngology, screening of 20000 asymptomatic individuals was performed using plasma Epstein Barr Virus DNA analysis. The presence of plasma EBV DNA consisting of short DNA fragments released by NPC cells helped identify NPC patients. In the published results, 34 NPC was identified in 300-screened positive individuals. In the rest of the cohort, NPC was not identified with initial nasoendoscopy and biopsy. A few more cancers was subsequently identified on Magnetic Resonance Imaging upon follow-up at 3 years and was confirmed with repeated endoscopic biopsies. In the current study the investigators would invite patients with persistently positive screening on plasma EBV-DNA analysis and no cancer found on usual diagnostic tests to undergo the novel screening endoscopy.

Individuals would be screened for eligibility at the clinic follow-up at the Department of Otorhinolaryngology. Study consent would be taken if they agree to participate in the current study.

Endoscopic procedures would be performed by endoscopists with expertise on performing magnifying NBI endoscopy at the Combined Endoscopy Center, Prince of Wales Hospital. It would be conducted at the Combined Endoscopy Center, Prince of Wales Hospital. Topical local anaesthetic will be applied to the oropharynx and nasopharynx. In addition, intravenous sedation by use of Midazolam and Fentanyl would be given. Endoscopes with magnification and NBI function would be used (GF-H290Z, Olympus Medical Corporations, Tokyo, Japan). A soft black hood would be attached to the tip of the endoscope for better focal length adjustment.

Upon insertion through a mouthpiece, the scope will then be retroflexed into the nasopharynx and the lateral walls into the Fossa of Rosenmuller and the posterior nasopharyngeal wall will be systematically examined with white light and NBI. Target suspicious areas would be examined by use of magnification with the power up to 80X. Biopsy would be taken if suspicious lesion is identified during the procedure.

In addition, non-contrast Magnetic Resonance Imaging (MRI) of the nasopharynx would be performed if the participants have not received a similar scan in recent 6 months and have no contra-indications to MRI. The MRI finding would be correlated with the endoscopic and histological findings.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥ 18 years old
2. Positive result on plasma EBV-DNA analysis
3. No cancer identified on conventional investigations including nasoendoscopy and MRI

Exclusion Criteria:

1. History of nasopharyngeal, oropharyngeal cancer
2. Patients on anticoagulation (Including warfarin and other direct oral anti-coagulants)
3. Bleeding tendency (International Normalized Ratio (INR) > 1.5 or Platelet < 50 x109/L)
4. Trismus, unable to pass oral endoscope
5. Allergic to local anaesthetic agents (Lignocaine)
6. Failure of vital organ (heart, lungs, liver, or kidneys) function
7. Other conditions deemed unsuitable for endoscopy
8. Refusal to participate, or inability to sign consent for study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Newly diagnosed Nasopharyngeal cancer | 1 month
  Newly diagnosed nasopharyngeal cancer with the novel endoscopic approach

SECONDARY OUTCOMES:
Rate of Adverse event - overall | 7 days
  Rate of Adverse event related to the endoscopic procedure
Rate of adverse event - haemorrhage | 7 days
  Rate of haemorrhage related to the endoscopic procedure
Rate of adverse event - perforation | 7 days
  Rate of perforation related to the endoscopic procedure
Rate of adverse event - infection | 7 days
  Rate of infection related to the endoscopic procedure
Rate of adverse event - aspiration pneumonia | 7 days
  Rate of aspiration pneumonia related to the endoscopic procedure
Stage of the newly diagnosed nasopharyngeal cancer | 1 month
  TNM stage distribution of the newly diagnosed NPC
Duration of the endoscopic procedure | 1 day
  Duration from scope insertion to scope withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, MBChB, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No